CLINICAL TRIAL: NCT03717545
Title: Second Transplantation for Graft Failure After First Allogeneic Stem Cell Transplantation
Brief Title: Second Transplantation for Graft Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaojun Huang,MD, Head of Peking University Institute of Hematology, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2nd tx for GF
Record Dates: First submitted 2018-09-30; First posted 2018-10-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Graft Failure; Stem Cell Transplant Complications

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention arm (Experimental): second allogeneic stem cell transplantation
  Interventions: Other: second allogeneic stem cell transplantation

INTERVENTIONS:
Other: second allogeneic stem cell transplantation — 1. Change another donor
  2. conditioning regimen: FLU/CY/anti-CD25 moAb

SUMMARY:
Graft failure is a lethal complication after allogeneic stem cell transplantation, which often need a salvage transplantation. However, the current outcome of second transplantation for graft failure is far from satisfactory. We performed a prospective single-arm study to investigate the safety and efficacy of a novel regimen.

ELIGIBILITY:
Inclusion Criteria:

* graft failure after first allogeneic stem cell transplantation
* no active infection or GVHD or severe organ dysfunction
* sign written informed consent

Exclusion Criteria:

* active infection, GVHD, organ failure
* expected life < 28 days

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
engraftment | 28 days after second transplantation
  Engraftment of neutrophils was defined as the first of 3 consecutive days when the absolute neutrophil count achieved 500/uL.

SECONDARY OUTCOMES:
TRM at 28 day | 28 days after second transplantation
  treatment-related mortality(TRM) was defined as death from any cause other than relapse.
TRM at 100d | day 100 after second transplant
  treatment-related mortality(TRM) was defined as death from any cause other than relapse.
Overall survival at 100d | day100 after second transplantation
  Overall survival at 100d

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun YQ, Wang Y, Wang FR, Yan CH, Cheng YF, Chen YH, Zhang YY, Han TT, Han W, Suo P, Xu LP, Zhang XH, Liu KY, Huang XJ. Graft Failure in Patients With Hematological Malignancies: A Successful Salvage With a Second Transplantation From a Different Haploidentical Donor. Front Med (Lausanne). 2021 Jun 4;8:604085. doi: 10.3389/fmed.2021.604085. eCollection 2021. PMID 34150785